CLINICAL TRIAL: NCT02718391
Title: Complementary Vaccination With Dendritic Cells Pulsed With Autologous Tumor Lysate in Resected Stage III and IV Melanoma Patients: a Phase II Randomized Trial (ACDC Adjuvant Trial)
Brief Title: Complementary Vaccination With Dendritic Cells Pulsed With Autologous Tumor Lysate in Resected Stage III and IV Melanoma Patients.
Acronym: ACDC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The randomization to the observational arm of the trial was no longer ethical
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST172.04; 2014-005123-27 (EudraCT Number)
Record Dates: First submitted 2016-01-21; First posted 2016-03-24 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2019-04

CONDITIONS: Malignant Melanoma; Adjuvant Drug Therapy; Vaccin Therapy
Keywords: Intradermal Autologous Dendritic Cell Vaccine; Malignant Melanoma; Adjuvant; vaccin; therapy; randomized trial; observation
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Autologous Dendritic Cell vaccine (Experimental): Daily 3 MU Interleukin 2 will be administered subcutaneously for 5 days starting from the second day after each vaccine dose. Vaccine doses will be given intradermally in two sites close to inguinal or axillary lymphnode stations that had not site of previous surgical exeresis.The first dose (WK1) will consist of freshly prepared vaccine, whereas for all the further doses cryopreserved aliquots will be utilized. The remaining 5 doses will be administered every 4 weeks to complete six months of therapy (six vaccines).
  Interventions: Biological: Autologous Dendritic Cell vaccine
- Arm B: follow up (No Intervention): Arm B: Patients will undergo laboratory and clinical assessment, tumor re-staging, blood collection for immunological biomarkers every 12 weeks until relapse.

INTERVENTIONS:
Biological: Autologous Dendritic Cell vaccine — The Dendritic Cells vaccine is given intradermally with 5 injections in sites close to inguinal or axillary lymphnode stations that had not site of previous surgical exeresis; as a rule, vaccine administrations should be performed by alternating injections sites. Two days after each vaccine administration, daily 3 MU Interleukin 2 will be administered subcutaneously for 5 days.
  Arms: Arm A: Autologous Dendritic Cell vaccine

SUMMARY:
This phase II, randomized, open-label trial aims to assess whether the vaccination increase RFS in disease free melanoma patients after surgery. Patients will be randomized between Intradermal Autologous Dendritic Cell Vaccine loaded with autologous tumor lysate or homogenate (6 vaccines every 4 weeks) and observation.

DETAILED DESCRIPTION:
This study will be a randomized phase II trial (1:1 allocation ratio) in resected stage III/IV melanoma patients. The randomization list will be stratified by stage (III and IV M1a-b and IVM1c), and time from primitive tumor to first metastasis (≤ 2 years versus > 2 years). Five randomization lists will be defined, one for each stratum.

On the basis of literature, the investigators assume a median relapse-free survival of 7.0 months for the standard group. With a two-sided tailed alpha of 0.10 and power of 80%, assuming a median relapse-free survival of 11.7 months in the experimental arm (hazard ratio 0.60), it will be necessary to recruit 60 patients per arm over a period of 24 months and to have a subsequent 12 months of follow-up. In the context of data monitoring board activities, an interim analysis for futility, according to the Bayesian approach, will be performed at 18 months in order to control the safety.

Primary endpoints will be relapse free survival. Secondary end points will be OS, In vivo and in vitro immunomonitoring. Immunologic efficacy will be measured by best Delayed Type Hypersensitivity score (reactivity to lysate or KLH) obtained after at least 4 vaccine doses, alone or combined with Interferon-g ELISPOT analysis of tumor antigen-specific circulating effectors obtained after a minimum of 4 vaccine doses, both compared with prevaccine samples. In vivo monitoring will focus on functional phenotyping of circulating immune effectors/regulators, functional characterization of circulating tumor antigen-specific immune effectors and regulators, and identification of serum markers that are predictive of response.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent: patients must be willing and able to give written informed consent, that have to be given before starting of screening procedure.
2. Availability of autologous tumor tissue fulfilling acceptance criteria prescribed by the "Product Specification File".
3. Patients must have histologically or cytologically confirmed melanoma (all type of melanomas);
4. Patients must be disease free after surgical removal of a metastatic lesions (stage IV or metachronous stage III)
5. Eastern Cooperative Oncology Group performance status 0-1
6. Negative screening tests for HIV, Hepatitis B virus, Hepatitis C virus and syphilis not older than 30 days before performing any of the Good Manufacturing Practice-regulated activities required (leukapheresis, collection of tumor biopsies to be used for tumor lysate/homogenate preparation);
7. Men and women aged ≥ 18 years.
8. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up 8 weeks after the study, in order to minimize the risk of pregnancy;
9. Patients must have normal organ and marrow function according to clinical practice.

Exclusion Criteria:

1. Patients who have positive tests to Hepatitis B virus, Hepatitis C virus HIV, or syphilis (specific blood testing must be performed within 30 days before any Good Manufacturing Practice-regulated activity (leukapheresis and collection of tumor biopsies to be used for tumor lysate preparation).
2. Patients who have had prior lines of systemic chemotherapy, immunotherapy or biological therapy for metastatic melanoma.
3. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements (on physician's judgment).
5. Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 3 years (except for previously treated basal cell carcinoma and in situ carcinoma of the uterine cervix);
6. Any contraindication to undergo leukapheresis as evaluated by transfusionist (e.g. severe anemia, thrombocytopenia, oral anticoagulant therapy) or to undergo surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | The time from the date of randomization to the date of the first relapse or the date of death from any cause or the date of the last restaging in non relapsed patients, assessed up to 36 months

SECONDARY OUTCOMES:
Overall survival (OS) | From the date of randomization until the date of death from any cause or the last date the patient was known to be alive, assessed up to 36 months
Immunologic efficacy will be measured by best delayed-type hypersensitivity score (reactivity to lysate or KLH) obtained after at least 4 vaccine doses | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ridolfi, MD, Principal Investigator — IRST IRCCS
Locations (2):
- Italy (2):
  - UO Immunoterapia e laboratorio TCS, IRST IRCCS, Meldola, FC
  - UO Oncologia Medica, IRCCS IRST, Meldola (FC), FC

REFERENCES:
- [Derived] Bulgarelli J, Piccinini C, Scarpi E, Gentili G, Renzi L, Carloni S, Limarzi F, Pancisi E, Granato AM, Petrini M, De Rosa F, Guidoboni M, Fanelli D, Tumedei MM, Tazzari M, Baravelli S, Bronico I, Cortesi P, Pignatta S, Capelli L, Ancarani V, Foschi G, Turci L, Tauceri F, Framarini M, Ridolfi L. Adjuvant dendritic cell-based immunotherapy in melanoma: insights into immune cell dynamics and clinical evidence from a phase II trial. J Transl Med. 2025 Apr 18;23(1):455. doi: 10.1186/s12967-025-06403-8. PMID 40251644